CLINICAL TRIAL: NCT05756283
Title: The PREHAAAB Trial: Multimodal Prehabilitation for Patients Awaiting Open Abdominal Aortic Aneurysm Repair - An International Randomized Controlled Trial
Brief Title: The PREHAAAB Trial: Multimodal Prehabilitation for Patients Awaiting Open Abdominal Aortic Aneurysm Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Heather Gill, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PREHAAAB Trial
Record Dates: First submitted 2023-02-14; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Prehabilitation; Exercise; Nutrition; Quality of life; Postoperative Complications; Psychosocial intervention
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Motor Activity; Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Prehabilitation (Experimental): Participants in the intervention group will undergo, in addition to the standard of care, 6+/-1 weeks of a personalized multimodal prehabilitation program. The interventions included will be patient-centered, aiming to optimize patients' preoperative health status while enhancing their empowerment and engagement.
  Interventions: Behavioral: Multimodal Prehabilitation
- Control group (standard of care) (No Intervention): Participants in the control group will receive the standard of care. This will include comorbidity optimization, anemia correction and smoking cessation advice if deemed appropriate.

INTERVENTIONS:
Behavioral: Multimodal Prehabilitation — EXERCISE
  * Supervised exercise
    * High intensity interval training
    * Strength exercise
  * Home-based exercise / promotion of physical activity
    * Low-moderate intensity aerobic training
    * Inspiratory muscle training
    * Low-moderate intensity strength training
  NUTRITION: nutrition education and optimization. Intake of 0.4g/kg of whey isolate after every supervised training.
  PSYCHOSOCIAL: mindfulness, cognitive reframing and coping strategies.
  Arms: Multimodal Prehabilitation

SUMMARY:
An abdominal aortic aneurysm is a condition where the major artery in the abdomen becomes larger than usual. Over time, as it continues to grow, the wall of the artery weakens and there is a risk that the artery can burst causing internal bleeding and death. Aortic aneurysms are fixed when they reach a certain size to prevent that outcome. The surgery to fix them is a major, high-risk surgery that is associated with a lot of complications and a slow recovery back to normal. The time between diagnosis and surgery is called the pre-operative period and is a key time to optimize a patient's health in order to ensure the best possible outcomes following surgery. This study will look at whether a multidisciplinary pre-operative program that involves exercise training, nutritional advice and supplementation, and psychosocial support will reduce complications following surgery. This program should decrease complications and speed up a patient's recovery back to normal after surgery. It is also a way for patients to take ownership of their disease and play an active role in their health care journey. The benefits from this program will go beyond the pre-operative time frame, as the habits and knowledge gained will improve their health over their lifetime. This study will also assess the economic impact and cost of a program like this.

DETAILED DESCRIPTION:
Abdominal aortic aneurysms (AAA) are asymptomatic until they rupture, which carries an 80- 90% mortality. Therefore, AAA are surgically repaired when they reach 5.0 cm in women and 5.5cm in men. Despite advances to surgical technique and peri-operative care, open surgical repair still carries a high incidence of post-operative complications of 30-40%, and a long recovery period. This is largely because the surgery itself is major abdominal surgery, and these patients often have significant comorbidities and low functional status. Multimodal prehabilitation (MP) is a concept that uses the preoperative timeframe (between diagnosis and surgery) to optimize physical, nutritional, and emotional wellbeing to improve a patient's functional status and ability to withstand the stress of surgery. To date, there is no study evaluating the effect of MP on post-operative complications following open AAA repair.

The primary objective of this trial is to determine if MP will decrease complications as measured by the comprehensive complication index following open AAA repair compared to standard of care. This trial will also assess the effect of MP on functional capacity, hospital length of stay, 30-day mortality and health related quality of life, as well as to assess cost effectiveness, adherence, and fidelity to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than 50 years of age awaiting elective open AAA repair with AAA diameter ≤6.9cm. Participants should have the ability to give informed consent.

Exclusion Criteria:

* Participants undergoing thoracic, thoracoabdominal and/or perivisceral AAA repair.
* Participants with ruptured or symptomatic AAA.
* Participants with AAA maximal diameter ≥7cm.
* Physical inability to exercise: severe osteoarthritis, musculoskeletal or neurological impairment that precludes exercise.
* Contraindication to exercise: rest systolic blood pressure ≥ 180 mmHg and/or diastolic ≥ 100 mmHg, uncontrolled atrial or ventricular arrythmias or proven exercise induced arrhythmias, unstable angina, unstable or acute heart failure, severe symptomatic valvular stenosis, dynamic left ventricular outflow tract obstruction or other comorbidities that imply clinical instability.
* Cognitive impairment that would impede understanding of study procedures, informed consent or study questionnaires or the inability to effectively communicate in English/French/Spanish/Catalan.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications measured by the Comprehensive Complication Index (CCI) | CCI will be measured from admission to 6 weeks postoperatively
  The CCI was developed to address some of the limitations of traditional surgical morbidity reporting, such as only reporting the most severe complication or only picking the most common types of complications. It is scored on a true linear interval scale from 0-100 and incorporates the totality of all complications and their severity experienced by a patient

SECONDARY OUTCOMES:
ICU Length of stay | From admission to 6 weeks postoperatively
  Intensive Care Unit length of stay
Hospital length of stay | From admission to 6 weeks postoperatively
  Days from admission to discharge from the hospital
Reinterventions | from surgery day to 6 week postoperatively
  Need for surgical reintervention due to surgical complications
Readmission | at 6 weeks and at 1 year postoperatively
  Readmission to the hospital
Emergency Room visits | at 6 weeks and at 1 year postoperatively
  Visits to the emergency room with or without admission to the hospital
6-Minute Walk Test | Measured at baseline, preoperatively and 6 weeks postoperatively
  6-minute walk test
VO2 peak | Measured at baseline and preoperatively
  Oxygen consumption at peak exercise
VO2 AT | Measured at baseline and preoperatively
  Oxygen consumption at anaerobic Threshold
VE/VCO2 | Measured at baseline and preoperatively
  Minute ventilation/carbon dioxide production
Yale physical activity survey (YPAS) | Measured at baseline, preoperatively, 6 weeks and 1 year postoperatively
  Questionnaire of daily physical activity
SF36 | Measured at baseline, preoperatively, 6 weeks and 1 year postoperatively
  Quality of life questionnaire
Depression | Measured at baseline, preoperatively, 6 weeks and 1 year postoperatively
  Depression measured by the Hospital Anxiety and Depression questionnaire (HADS) 0 (no depression)- 21 (maximal depression)
Anxiety | Measured at baseline, preoperatively, 6 weeks and 1 year postoperatively
  Anxiety measured by the Hospital Anxiety and Depression questionnaire (HADS) 0 (no anxiety)- 21 (maximal anxiety)
Patient Generated Subjective Global Assessment (PG-SGA) | Measured at baseline, preoperatively
  Malnutrition assessment tool
Compliance to intervention | Measured from baseline to preoperatively
  Compliance to the different components of the intervention, measured by attendance to supervised sessions (%), adherence to nutritional counseling and supplementation (%), adherence to home-based exercise (%) and adherence to the psychosocial sessions (%)
Fidelity to exercise intervention | Measured from baseline to preoperatively
  Real training wattage and kg vs expected
Height | Measured at baseline and preoperatively
  measurement of height in meters
Weight | Measured at baseline and preoperatively
  measurement of Weight in kg
Body Mass Index (BMI) | Measured at baseline and preoperatively
  Measurement of body mass index (weight and height will be combined to report BMI in kg/m^2)
Body Fat percentage | Measured at baseline and preoperatively
  Measurement of body fat percentage using Bioelectrical Impedance Analysis
Fat Free Mass (FFM) | Measured at baseline and preoperatively
  Measurement of body fa free mass in kg, using Bioelectrical Impedance Analysis
Muscle Mass | Measured at baseline and preoperatively
  Measurement of muscle mass in kg, using Bioelectrical Impedance Analysis
Phase angle | Measured at baseline and preoperatively
  Measurement of phase angle, using Bioelectrical Impedance Analysis
Satisfaction and acceptability | Preoperative assessment
  Intervention satisfaction and acceptability questionnaire
Incidents of adverse events (prehabilitation safety and tolerability) | Measured from Baseline to Preoperatively
  Incidence of adverse events and severe adverse events during prehabilitation program
Quality adjusted life years | Measured at baseline, preoperatively, 6 weeks and 1 year postoperatively
  Quality adjusted life years derived from SF36 data (SF6D)
Prehabilitation cost-effectiveness | Measured at 1 year postoperatively
  Measurement of prehabilitation cost-effectiveness using data from SF6D, prehabilitation costs and hospitalization related costs.

CONTACTS AND LOCATIONS:
Locations (1):
- MUHC-RIMUHC Royal Victoria Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Barakat HM, Shahin Y, Khan JA, McCollum PT, Chetter IC. Preoperative Supervised Exercise Improves Outcomes After Elective Abdominal Aortic Aneurysm Repair: A Randomized Controlled Trial. Ann Surg. 2016 Jul;264(1):47-53. doi: 10.1097/SLA.0000000000001609. PMID 26756766
- [Background] Tew GA, Batterham AM, Colling K, Gray J, Kerr K, Kothmann E, Nawaz S, Weston M, Yates D, Danjoux G. Randomized feasibility trial of high-intensity interval training before elective abdominal aortic aneurysm repair. Br J Surg. 2017 Dec;104(13):1791-1801. doi: 10.1002/bjs.10669. Epub 2017 Oct 9. PMID 28990651
- [Background] Fenton C, Tan AR, Abaraogu UO, McCaslin JE. Prehabilitation exercise therapy before elective abdominal aortic aneurysm repair. Cochrane Database Syst Rev. 2021 Jul 8;7(7):CD013662. doi: 10.1002/14651858.CD013662.pub2. PMID 34236703
- [Background] Staiger RD, Cimino M, Javed A, Biondo S, Fondevila C, Perinel J, Aragao AC, Torzilli G, Wolfgang C, Adham M, Pinto-Marques H, Dutkowski P, Puhan MA, Clavien PA. The Comprehensive Complication Index (CCI(R)) is a Novel Cost Assessment Tool for Surgical Procedures. Ann Surg. 2018 Nov;268(5):784-791. doi: 10.1097/SLA.0000000000002902. PMID 30272585
- [Derived] Coca-Martinez M, Doonan RJ, Gillis C, Mackenzie K, Obrand DI, Bayne JP, Steinmetz OK, Girsowicz E, Lopez-Baamonde M, Jessula S, Yugueros X, Martinez-Palli G, Gill HL. The PREHAAAB Trial: Multimodal prehabilitation for patients awaiting open abdominal aortic aneurysm repair - A study protocol for an international randomized controlled trial. PLoS One. 2025 Dec 29;20(12):e0339473. doi: 10.1371/journal.pone.0339473. eCollection 2025. PMID 41460856